CLINICAL TRIAL: NCT05777525
Title: Use of Essential Oils as Natural Therapies Against Dermatophytosis and New Diagnostic Techniques
Brief Title: Use of Essential Oils as Natural Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Ana María Pérez Pico, Clinical Professor, University of Extremadura
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CreamAAT
Record Dates: First submitted 2023-02-13; First posted 2023-03-21 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Dermatophytoses; Skin Lesion
Keywords: Echography; essential oils; dermatophytosis; natural treatment; ultrasonography
MeSH Terms: conditions — Tinea

STUDY DESIGN:
Intervention Model Description: Parallel treatment design and double-blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Echography (No Intervention): Ultrasound skin measurements will be taken before and after the enriched cream treatment.
- "Visiopor PP-34 camera" (No Intervention): Measurements of the skin will be taken by "Visiopor PP-34" camera before and after the treatment with enriched cream.
- Mycological culture (No Intervention): Skin samples will be taken and analyzed by mycological culture before and after treatment with enriched cream
- treatment application (Experimental): The essential oil enriched cream will be applied to study participants.
  Interventions: Combination Product: application of cream "La Chinata"

INTERVENTIONS:
Combination Product: application of cream "La Chinata" — application of cream enriched with essential oil
  Arms: treatment application

SUMMARY:
Mycosis is defined as a fungal infection caused by the implantation of etiological agents that compromises the dermis and subcutaneous tissue.

Dermatophytosis is a fungal infection caused by dermatophytes, being the main cause of superficial mycoses and constituting an important public health problem.

The production or development of infections is due in any case to the loss of ability to protect the exterior of the skin epidermis and, in the case of nails, to the fact that the nail apparatus does not have cell-mediated immunity effective, thus being more susceptible to infection than other parts of the skin. Although these infections can be bacterial, fungal, or viral, the investigators will focus on fungal infections.

There are numerous studies that suggest the suitability of EOs as an alternative treatment for fungal infections.

Due to this, in this project the investigators will analyze one of the most important infections within the podiatric health of the population, in terms of its incidence, pathogenesis, diagnostic methods, etc., and for this our research will be focused on examining whether there is improvements in the skin of patients with dermatophytosis treated with cream enriched with natural oils, in our case tea tree oil, verified by ultrasound.

DETAILED DESCRIPTION:
Mycosis is defined as a fungal infection caused by the implantation of etiological agents that compromise the dermis and subcutaneous tissue. The etiological agents can be filamentous fungi, yeasts and mold fungi, present in nature, in the soil, vegetation and in decomposing organic matter. Mycosis is among the most common form of infection in humans, with an approximate incidence of 20-25% of the world population.

Dermatophytosis is the fungal infection caused by dermatophytes, being the main cause of superficial mycoses and constituting an important public health problem. Dermatophytes are divided into three genera, having an affinity for and the ability to grow in keratinized tissues, such as hair, skin, and nails. Other fungal infections of the skin and appendages in humans may be caused by non-dermatophyte fungi, such as yeasts and mold fungi. Onychomycosis is dermatophytosis that affects the nails, this being one of the most frequent causes in the clinic, both in the dermatological field and in general medicine. In this type of infections, the most important thing is to know the agent that causes the infection, thus being able to establish a specific treatment. Currently, approximately 90% of toenail onychomycosis and 75% of all nail onychomycosis are caused by dermatophytes. The production or development of infections is due in any case to the loss of ability to protect the exterior of the skin epidermis and, in the case of nails, to the fact that the nail apparatus does not have cell-mediated immunity effective, thus being more susceptible to infection than other parts of the skin. Although these infections can be bacterial, fungal, or viral, the investigators will focus on fungal infections.

Various scientific articles have verified and confirmed that superficial fungal infection (tinea pedis, athlete's foot, tinea versicolor, etc.) is usually referred to the foot, due to its transmission through showers and shared materials, environmental humidity , etc.

There are numerous studies that suggest the suitability of EOs as an alternative treatment for fungal infections and the investigators found numerous studies that demonstrate the antifungal action of various commercial EOs in in vitro studies. Among the most studied EOs due to their antifungal activity, the following stand out: thyme (Thymus vulgaris), cinnamon (Cinnamomun zeylanicum) and tea tree (Melaleuca alternifolia), among many others.

Due to this, in this project we will analyze one of the most important infections within the podiatric health of the population, in terms of its incidence, pathogenesis, diagnostic methods, etc., and for this our research will be focused on examining whether there is improvements in the skin of patients with dermatophytosis treated with cream enriched with natural oils, in our case tea tree oil, verified by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* who is in the age range
* consent signature accepted
* not have allergies to the treatment
* not have chronic skin diseases

Exclusion Criteria:

* not meet any inclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Appearance of the skin through the use of ultraviolet light through the processing of photographs obtained | 3 months
  Data collection with Visiopor camera. Measurement unit: occupied area
Skin thickness measured in millimeters through images obtained by ultrasound | 3 months
  Data collection with ultrasound. Measurement unit: millimeters
Taking mycological samples for subsequent cultivation on saboureaud agar | 3 months
  take mycological samples to check for infection. Measurement unit: positive/negative

CONTACTS AND LOCATIONS:
Locations (1):
- Raquel Mayordomo Acevedo, Plasencia, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT05777525/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05777525/ICF_001.pdf